CLINICAL TRIAL: NCT00092963
Title: A Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Examine the Efficacy of Rizatriptan 10 mg Tablet Administered Early During a Migraine Attack While the Pain is Mild
Brief Title: Study to Test an Approved Product in the Early Treatment of Migraine (0462-065)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-065; 2004_022
Record Dates: First submitted 2004-09-28; First posted 2004-09-29 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0462, rizatriptan benzoate / Duration of Treatment: 1day
Drug: Comparator: placebo / Duration of Treatment: 1 day

SUMMARY:
The purpose of this study is to test the effectiveness of an approved drug in the early treatment of migraine while the pain is still mild.

ELIGIBILITY:
Inclusion Criteria:

* 6-month history of migraine
* Migraine attacks typically mild when they begin with 1-4 migraine attacks per month

Exclusion Criteria:

* Heart disease
* High blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2004-08-17 (Actual); Primary Completion 2005-01-14 (Actual); Study Completion 2005-01-14 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who are pain free at 2 hours postdose.
Tolerability as measured by subjective adverse experience reporting.

SECONDARY OUTCOMES:
Percentage of patients with 24 hour sustained pain freedom
Percentage of patients free at 30/45/60/90 minutes postdose
Percentage of patients with associated symptoms at 2 hours
Percentage of patients requiring rescue med between 2 & 24 hours
Percentage of patients with functional disability at 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Cady R, Martin V, Mauskop A, Rodgers A, Hustad CM, Ramsey KE, Skobieranda F. Efficacy of Rizatriptan 10 mg administered early in a migraine attack. Headache. 2006 Jun;46(6):914-24. doi: 10.1111/j.1526-4610.2006.00466.x. PMID 16732837
- [Background] Martin V, Cady R, Mauskop A, Seidman LS, Rodgers A, Hustad CM, Ramsey KE, Skobieranda F. Efficacy of rizatriptan for menstrual migraine in an early intervention model: a prospective subgroup analysis of the rizatriptan TAME (Treat A Migraine Early) studies. Headache. 2008 Feb;48(2):226-35. doi: 10.1111/j.1526-4610.2007.00947.x. Epub 2007 Nov 13. PMID 18005144
- [Background] Cady R, Martin V, Mauskop A, Rodgers A, Hustad C, Ramsey K, Skobieranda F. Symptoms of cutaneous sensitivity pre-treatment and post-treatment: results from the rizatriptan TAME studies. Cephalalgia. 2007 Sep;27(9):1055-60. doi: 10.1111/j.1468-2982.2007.01391.x. Epub 2007 Aug 6. PMID 17681023
- [Background] Ho TW, Rodgers A, Bigal ME. Impact of recent prior opioid use on rizatriptan efficacy. A post hoc pooled analysis. Headache. 2009 Mar;49(3):395-403. doi: 10.1111/j.1526-4610.2009.01346.x. Epub 2008 Feb 12. PMID 19222588